CLINICAL TRIAL: NCT06067698
Title: Clinical Study Evaluating the Efficacy and Safety of Alpha-lipoic Acid in Patients With Ulcerative Colitis Treated With Mesalamine
Brief Title: Alpha Lipoic Acid in Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Farouk, Clinical pharmacy manager, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36264MS206/6/23
Record Dates: First submitted 2023-09-15; First posted 2023-10-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (Placebo) (Placebo Comparator): (Placepo group; n=30) which will receive mesalamine 1000 mg three times daily plus placebo once daily
  Interventions: Drug: "Mesalamine" and "Placebo"
- Group (Alpha lipoic acid) (Active Comparator): (Alpha-lipoic acid group; n=30) which will receive mesalamine 1000 mg three times daily plus alpha-lipoic acid 600 mg
  Interventions: Drug: "Mesalamine" and "alpha-lipoic acid"

INTERVENTIONS:
Drug: "Mesalamine" and "alpha-lipoic acid" — Mesalamine 1000 mg every 8 hrs. + alpha-lipoic acid 600 mg once daily for 3 months
  Arms: Group (Alpha lipoic acid)
Drug: "Mesalamine" and "Placebo" — Mesalamine 1000 mg every 8 hrs. + Placebo once daily for 3 months
  Arms: Group (Placebo)

SUMMARY:
This study aims at evaluating the efficacy and safety of alpha-lipoic acid as adjuvant therapy to mesalamine in patients with mild to moderate ulcerative colitis due to its effect as anti-oxidant and anti-inflammatory drug which can help to improve disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both male and female sex.
* Newly diagnosed patients with active mild and moderate ulcerative colitis according to American College of Gastroenterology (ACG) Clinical Guideline for diagnosing Ulcerative Colitis in Adults.26
* Patients treated with 5-aminosalisylic acid (mesalamine).

Exclusion Criteria:

* Patients with severe ulcerative colitis.
* Patients with colorectal cancer.
* Patients on rectal or systemic steroids.
* Patients on immunosuppressants or biological therapies.
* Patients with previously failed treatment with sulphasalazine.
* Patients with known allergy to study medications.
* History of complete or partial colectomy.
* Patients with significant liver disease (fibrosis, cirrhosis, NASH, NAFLD).
* Patients with other inflammatory diseases.
* Patients with thyroid diseases.
* Patients with arrhythmia, ischemic heart disease, and heart failure.
* Patients with diabetes.
* Patients on antioxidants supplement (vitamin A, C, E), selenium, co-enzyme Q.
* Patients on amlodipine, levothyroxine, low strength aspirin, warfarin, atorvastatin, insulin, oral hypoglycemic, chemotherapy (drug-drug interaction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in both health related quality of life | 3 months from start of treatment
  The Short Inflammatory Bowel Disease Questionnaire to evaluate quality of life to the patient through score from 1 to 7 whether higher scores mean a better outcome and lower score mean a worse outcome
Change in disease severity | 3 months from start of treatment
  Partial Mayo Scoring Index which evaluate severity through total score whether higher scores mean a worse and lower score mean a better outcome.

SECONDARY OUTCOMES:
Change in "fecal calprotectin" as biological parameters | 3 months from start of treatment
  measure Fecal calprotectin which lower result means a better outcome
Change in "reduced glutathione" as biological parameters | 3 months from start of treatment
  measure reduced glutathione which lower result means a better outcome
Change in "interleukin-6" as biological parameters | 3 months from start of treatment
  measure interleukin-6 which lower result mean better outcome.
Change in "Transforming growth factor - beta 1" as biological parameters | 3 months from start of treatment
  measure Transforming growth factor - beta 1 which lower result mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanat university hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No